CLINICAL TRIAL: NCT01602133
Title: A Clinical Assessment of an Ultrasound-guided Inserted Peripheral Intravenous Catheter
Brief Title: Assessment of Ultrasound-guided Inserted Peripheral Intravenous Catheter
Acronym: ECLIPSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prodimed SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2011-A01570-41
Record Dates: First submitted 2012-05-17; First posted 2012-05-18 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Venous Puncture
Keywords: venous puncture; seldinger technique; ultrasound guidance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- one intervention arm (Experimental)
  Interventions: Procedure: peripheral venous puncture

INTERVENTIONS:
Procedure: peripheral venous puncture — Ultrasound imaging of the arm is performed. If a suitable vein is identified, a percutaneous puncture is performed under ultrasound guidance. Then, an intravenous catheter is inserted according Seldinger method.

SUMMARY:
Evaluate the safety and efficacy of an an ultrasound-guided inserted peripheral intravenous catheter during a period of seven days.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with need of an intravenous therapy on peripheral line
* Unsuccessful attempts at establishing a peripheral intravenous line by nurse
* Age over 18 YO
* Written informed consent obtained

Exclusion Criteria:

* pregnant woman
* local contra-indication for venous puncture
* unconscious patient
* need of intravenous therapy requiring central line

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
length of use of the catheter measured in number of days | seven days

SECONDARY OUTCOMES:
adverse event during the period of use of the catheter | seven days
  extravasation and/or catheter removal before the end of the treatment and/or local complications (bleeding, neurologic trouble, venous thrombosis..)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Meyer, MD, Principal Investigator — Centre Hospitalier Sud Francilien- Corbeil- France
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

REFERENCES:
- [Derived] Tada M, Yamada N, Matsumoto T, Takeda C, Furukawa TA, Watanabe N. Ultrasound guidance versus landmark method for peripheral venous cannulation in adults. Cochrane Database Syst Rev. 2022 Dec 12;12(12):CD013434. doi: 10.1002/14651858.CD013434.pub2. PMID 36507736